CLINICAL TRIAL: NCT06254560
Title: The Study of Rituximab in the Treatment of Severe Aplastic Anemia With Platelet Transfusion Refractoriness
Brief Title: Rituximab for Serious Aplastic Anemia With Platelet Transfusion Refractoriness
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023NCRCA0113
Record Dates: First submitted 2024-01-19; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-02

CONDITIONS: Severe Aplastic Anemia; Platelet Transfusion Refractoriness
Keywords: Severe aplastic anemia; Platelet transfusion refractoriness; Rituximab
MeSH Terms: conditions — Anemia, Aplastic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rituximab group (Experimental): Rituximab combined with cyclosporine
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab is administered at a dose of 100mg per week, a total of 4 times. Cyclosporin is administered at a dose of 3-5mg/kg per day.
  Other Names: Mabthera

SUMMARY:
Due to long-term dependence on platelet transfusion, some severe aplastic anemia (SAA) patients suffer platelet transfusion refractoriness (PTR). Unlike immune thrombocytopenia (ITP), glucocorticoids and human immunoglobulin (IVIg) are generally ineffective for PTR. Due to the lack of effective intervention methods, patients with PTR suffer increased platelet transfusions, bleeding events and treatment costs, prolonged hospital stays, and decreased survival rate. SAA with PTR has become a challenge for physicians. The experiment aims to explore the efficacy of rituximab in the treatment of SAA with PTR, and establish a new effective, safe treatment method with relatively low treatment cost.

DETAILED DESCRIPTION:
During the treatment period, Rituximab is administered at a dose of 100mg per week, a total of 4 times.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosed SAA with PTR
* Age>18 years old, regardless of gender
* Initial diagnosed SAA with PTR
* Age>18 years old, regardless of gender

Exclusion Criteria:

* Allergy to rituximab
* Severe active infection
* Hypogammaglobulinemia
* Pregnant and lactating women
* Heart failure (NYHA classification IV)
* Individuals with epilepsy, dementia, and other mental disorders that require medication treatment who cannot understand or follow the research protocol
* Chronic infections or other chronic diseases that may be risk to the experiment
* The researchers believe that it is not suitable for participants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The response and complete remission rate with Rituximab protocol. | 6 months
  Response will be evaluated at each clinic visit. Complete response (CR) was defined as achieving all three peripheral blood count criteria: (1) Hb level up to the normal range; (2) ANC≥1.5×109/L; (3) PLT≥100×109/L. Partial response (PR) was defined as transfusion independent, no longer meeting criteria for severe disease. Persistence of transfusion requirement or death was evidence of no response (NR).

SECONDARY OUTCOMES:
Relapse rate | 12 months and 60 months
  Relapse was defined as a responder who met criteria for SAA again after achieving response and keeping stable blood counts for at least 3 months.
Sustained response (SR) | 12 months and 60 months
  SR was defined as Hb > 10 g/dL at 12 months and 60 months, in the absence of any treatment.
Survival | 60 months
  Survival rate within 5 years after diagnosis
Clonal evolution to myelodysplasia and acute leukemia. | 60 months
  Clonal evolution within 5 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Huang Jinbo, MD., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Killick SB, Bown N, Cavenagh J, Dokal I, Foukaneli T, Hill A, Hillmen P, Ireland R, Kulasekararaj A, Mufti G, Snowden JA, Samarasinghe S, Wood A, Marsh JC; British Society for Standards in Haematology. Guidelines for the diagnosis and management of adult aplastic anaemia. Br J Haematol. 2016 Jan;172(2):187-207. doi: 10.1111/bjh.13853. Epub 2015 Nov 16. No abstract available. PMID 26568159
- [Background] Chockalingam P, Sacher RA. Management of patients refractory to platelet transfusion. J Infus Nurs. 2007 Jul-Aug;30(4):220-5. doi: 10.1097/01.NAN.0000281531.97183.c0. PMID 17667077
- [Background] Kerkhoffs JL, Eikenboom JC, van de Watering LM, van Wordragen-Vlaswinkel RJ, Wijermans PW, Brand A. The clinical impact of platelet refractoriness: correlation with bleeding and survival. Transfusion. 2008 Sep;48(9):1959-65. doi: 10.1111/j.1537-2995.2008.01799.x. Epub 2008 Jun 28. PMID 18564396